CLINICAL TRIAL: NCT05669833
Title: Guselkumab vs Golimumab in PsA TNF Inadequate Responder Patients: a Pragmatic Trial (EVOLUTION)
Brief Title: Guselkumab vs Golimumab in PsA TNF Inadequate Responder Patients
Acronym: EVOLUTION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1959PSA3006
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guselkumab 100mg q4w (Experimental): Guselkumab (GUS) 100mg every 4 weeks
  Interventions: Drug: Guselkumab
- Guselkumab 100mg q8w (Experimental): Guselkumab (GUS) 100mg every 8 weeks
  Interventions: Drug: Guselkumab
- Golimumab 50mg q4w (Active Comparator): Golimumab (GOL) 50mg every 4 weeks
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab (GUS) subcutaneous injection
  Other Names: Tremfya
  Arms: Guselkumab 100mg q4w; Guselkumab 100mg q8w
Drug: Golimumab — Golimumab (GOL) subcutaneous injection
  Other Names: Simponi
  Arms: Golimumab 50mg q4w

SUMMARY:
The trial is an open-label randomized study that will examine whether switching to a selective IL23 inhibitor (guselkumab) is more effective than switching to a second TNFi (golimumab) among patients with PsA who have an inadequate response to a TNFi.

DETAILED DESCRIPTION:
The primary aim of the trial will be to determine, among psoriatic arthritis (PsA) patients with an inadequate response (IR) to a tumor necrosis factor inhibitor (TNFi), whether switching to a new mechanism of action (MOA), specifically guselkumab (GUS), a selective interleukin 23 inhibitor (IL23i) targeting the p19 subunit, is more effective than switching to another TNFi. The primary hypothesis of this study is that switching to a new MOA may be more effective than switching to a second TNFi. This will be the first trial to test such a switch in PsA patients. Additionally, the proposed study will address the effectiveness of a new therapy, GUS, in a clinical practice setting among patients who are TNF IR.

ELIGIBILITY:
Inclusion Criteria:

1. Psoriatic arthritis meeting CASPAR criteria;
2. Active psoriatic arthritis defined by at least 1 swollen joint;
3. cDAPSA score ≥ 10; See also Exclusion #4 - cDAPSA must be > 14 in patients without psoriasis.
4. Using a TNFi or previously used a single TNFi historically and either never responded or lost response (TNF IR) and planning to switch to a new biologic therapy;
5. If using an oral small molecule/csDMARD (i.e., methotrexate, leflunomide, hydroxychloroquine, sulfasalazine, or apremilast), must be on a stable dose for 4 weeks and remain on a stable dose during the study; Use of up to two OSM/csDMARDs is allowed.
6. If using NSAIDs, glucocorticoids (<10 mg daily) or topical medications for psoriasis, must be on a stable dose for 4 weeks prior to Screening/Baseline 1 and remain on a stable dose during the study;
7. Age 18-80 (patients older than 80 may be more likely to have concomitant osteoarthritis which may make it difficult to assess whether symptoms are related to PsA vs OA).

Exclusion Criteria:

1. Prior exposure to golimumab or another non-TNFi biologic (IL12/23i, JAKi, an IL17i, or an IL23i); prior exposure to a TYK2i is acceptable, but cannot be used during course of the study;
2. An adverse event that precludes use of another TNFi (development of drug-induced SLE, allergic reaction, serious infection, heart failure symptoms, demyelination at any point during use of therapy) or any other contraindication or substantial intolerance to a TNFi;
3. Use of moderate to high dose glucocorticoids (>10 mg);
4. Already meets the primary endpoint at Baseline; [cDAPSA low disease activity ≤ 14; IGA of psoriasis 0/1] In patients with psoriasis, cDAPSA can be 10-14 IF the Investigator Global Assessment of Psoriasis ≥ 2.

   In patients without psoriasis, cDAPSA must be > 14 to meet eligibility requirements.
5. Currently pregnant or actively trying to conceive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Achievement of cDAPSA low disease activity | 12 Months
  Clinical Disease Activity in Psoriatic Arthritis (cDAPSA): a combination score of tender joint count, swollen joint count, patient assessment of pain, and patient global assessment of disease activity. Scale from 0-154 where higher figures indicate worse status. Remission is considered ≤4 and low disease activity >4 to ≤13.
Investigator Global Assessment of Psoriasis of Clear or Almost Clear | 12 Months
  Investigator global assessment (IGA) of psoriasis. A scale of 0-4 where higher figures indicate worse status. (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).

SECONDARY OUTCOMES:
Minimal Disease Activity (MDA) using PSAID-12 | 6 and 12 months
  Minimal Disease Activity (MDA) defines a satisfactory state of disease activity that includes 5 domains of PsA. 5/7 of the following criteria must be satisfied for MDA: patient global ≤ 2 (0-10), patient pain ≤ 2 (0-10), PSAID-12 <4 (0-10), TJC (Tender Joint Count) ≤ 1, SJC (Swollen Joint Count) ≤ 1, BSA (Body Surface Area) ≤ 3, and Leeds Enthesitis Index ≤ 1.
Minimal Disease Activity (MDA) using HAQ-DI | 6 and 12 months
  (MDA) Minimal Disease Activity defines a satisfactory state of disease activity that includes 5 domains of PsA. Participant would need to achieve 5/7 of the following criteria: patient global ≤ 2 (0-10), patient pain ≤ 2 (0-10), HAQ-DI (Health Assessment Questionnaire Disability Index) < 0.5 (0-3), TJC (Tender Joint Count) ≤ 1, SJC (Swollen Joint Count) ≤ 1, BSA (Body Surface Area) ≤ 3, and Leeds Enthesitis Index ≤ 1.
Change in PSAID-12 | 6 and 12 months
  Psoriatic Arthritis Impact of Disease Questionnaire 12-item questionnaire (PSAID-12) Survey. The range of the final PsAID-12 value is 0-10 where higher figures indicate worse status. Negative changes from baseline indicate improvement in disease activity.
PSAID-12 < 4 | 6 and 12 months
  Psoriatic Arthritis Impact of Disease Questionnaire 12-item questionnaire (PSAID-12) Survey. The range of the final PsAID-12 value is 0-10 where higher figures indicate worse status.
Change in DLQI | 6 and 12 months
  Dermatology Life Quality Index (DLQI) is a measure of skin disease activity. Calculated score of 0-30 where higher figures indicate worse status.Negative changes from baseline indicate improvement in disease activity.
IGA Among Patients with BSA > 3% at Baseline | 6 and 12 months
  Investigator global assessment (IGA) of psoriasis among patients with BSA (Body Surface Area) >3% at baseline. A scale of 0-4 where higher figures indicate worse status. (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
IGA Among Patients with IGA ≥ 2 at Baseline | 6 and 12 months
  Investigator global assessment (IGA) of psoriasis among patients with IGA of 2 or more (≥ 2) at baseline. A scale of 0-4 where higher figures indicate worse status. (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
Change in Promis Fatigue | 6 and 12 Months
  Promis Fatigue is a measure of fatigue with a score from 8-40 where higher figures indicate worse status. A negative change indicates less overall fatigue.
Resolution of Dactylitis | 6 and 12 Months
  Dactylitis is assessed using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. These results are summed to produce a final score ranging from 0 to 20. A higher score indicates more severe dactylitis. Resolution of dactylitis is defined as a dactylitis score of 0 with a baseline dactylitis score >0.
Resolution of Enthesitis | 6 and 12 Months
  Enthesitis is assessed using the Leeds Enthesitis Index (LEI). This measure includes the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The total LEI score of 0-6 is based on evaluating each of these six sites as 0 or 1 based on the absence or presence of pain/tenderness. Resolution of enthesitis is defined as a enthesitis score of 0 with a baseline enthesitis score >0.
Change in BASDAI | 6 and 12 Months
  Change in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) among patients with axial disease. The BASDAI sum score ranges from 0 to 10 and higher values indicate more active disease. Negative changes from baseline indicate improvement in disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (14):
- United States (14):
  - Family Arthritis Center, Loxahatchee Groves, Florida
  - Healing Rheumatology, Plant City, Florida
  - Southwest Florida Rheumatology, Riverview, Florida
  - Parris and Associates, Lilburn, Georgia
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University, New York, New York
  - Cincy Arthritis, Blue Ash, Ohio
  - Southern Ohio Rheumatology, Wheelersburg, Ohio
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Cumberland Rheumatology, Crossville, Tennessee
  - Heritage Rheumatology and Arthritis Care, Colleyville, Texas
  - Texas Arthritis Center, El Paso, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogdie A, Reddy SM, Gillespie SH, Husni ME, Scher JU, Salomon-Escoto K, Kay J, Luedders BA, Curtis JR, Shields AJS, Chakravarty SD, Gong C, Walsh JA. Guselkumab versus golimumab in patients with active psoriatic arthritis and inadequate response to an initial tumor necrosis factor inhibitor: study protocol for EVOLUTION, a pragmatic, phase 3b, open-label, randomized, controlled effectiveness trial. Trials. 2025 Mar 19;26(1):96. doi: 10.1186/s13063-025-08777-y. PMID 40102973